CLINICAL TRIAL: NCT04797806
Title: Phase III Study Comparing Anlotinib Plus Icotinib to Icotinib in Patients With Untreated Non-squmous NSCLC Harboring EGFR Concomitant Mutations
Brief Title: Study of Anlotinib Combined With Icotinib as the First-line Treatment in Patients With EGFR Concomitant Mutation NSCLC
Acronym: SAINT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SAINT
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-01

CONDITIONS: Non Small Cell Lung Cancer
Keywords: sensitive EGFR mutations and concomitant orthers; anlotinib; icotinib; first line; non-squamous NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib; icotinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combination therapy (Experimental): Anlotinib Combined With Icotinib
  Interventions: Drug: Anlotinib; Drug: Icotinib
- monotherapy (Other): Icotinib
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Anlotinib — Anlotinib 12 mg once a day from day 1 to 14 of a 21-day cycle.
  Arms: combination therapy
Drug: Icotinib — Icotinib：125 mg/tablet，three times a day，fasting or serving with food. It should be continued until disease progression or intolerable toxicity or patients withdraw of consent.

SUMMARY:
Evaluate the efficacy and safety of Anlotinib plus Icotinib as the first-line treatment in patients with sensitive EGFR concomitant mutations advanced non-small cell lung cancer

DETAILED DESCRIPTION:
Anlotinib Hydrochloride is a kind of innovative medicines approved by State Food and Drug Administration（CFDA:2011L00661） which was developed by Jiangsu Chia-tai Tianqing Pharmaceutical Co., Ltd. Anlotinib is a kinase inhibitor of receptor tyrosine with multi-targets, especially for VEGFR1、VEGFR2、VEGFR3、FGFR1/2/3、PDGFRa/β c-Kit and MET.

ELIGIBILITY:
Inclusion Criteria:

Signed and dated informed consent 18-75years，ECOG PS：0-2，Life expectancy of more than 3 months，with measurable lesion ( RECIST1.1) Histologically or cytologically confirmed, locally advanced and/or metastatic IIIB, IIIC or IV non-squamous NSCLC or recurrent non-squamous NSCLC（according to the 8th Edition of the AJCC Staging system）with EGFR 19 del or 21 L858R gene mutation and concomitant others.

Has not received chemotherapy or other targeted therapies；For recurrent disease, adjuvant chemotherapy, neoadjuvant chemotherapy or neoadjuvant chemotherapy plus adjuvant chemotherapy may be accepted, but recurrence occurs after ≥6 months from stopping treatment.

≥1 target lesion that has not received radiotherapy in the past 3 months and can be accurately measured in at least 1 direction；Previously received radiation therapy, but the radiotherapy area must be <25% of the bone marrow area, and radiation therapy must have closed for at least≥4 weeks at the time of enrollment; Main organs function is normal Patients of brain metastases with asymptomatic or mild symptoms can be enrolled The woman patients of childbearing age must agree to take contraceptive methods during the research and within another 8 weeks after treatment. Pregnancy test (blood serum test or urine) should be done within 7 days before the research and the result should be negative.The man patients who must agree to take contraceptive methods during the research and within another 8 weeks after treatment.

Exclusion Criteria:

Squamous cell carcinoma (including adenosquamous carcinoma); Small Cell Lung Cancer (including small cell cancer and other kinds of cancer mixed with non-small cell cancer) ALK-positive NSCLC Central Lung tumors that Imaging (CT or MRI) shows tumor lesions invade local large blood vessels; or with significant pulmonary cavum or necrotizing Patients with obvious brain metastases, cancerous meningitis, spinal cord compression, or with brain or pia mater disease. (patient with brain metastases who have completed treatment 14 days before and the symptoms are stable can be Enrolled, also should have no cerebral hemorrhage symptoms confirmed by brain MRI, CT or venography evaluation The patient is participating in other clinical studies or Participated in other anti-tumor drug clinical trials within 4 weeks before enrollment With other active malignancies that require simultaneous treatment Has a history of malignant tumors. Except for patients with cutaneous basal cell carcinoma, superficial bladder cancer, cutaneous squamous cell carcinoma or orthotopic cervical cancer who have undergone curative treatment and have no disease recurrence within 5 years after the start of treatment Patients with adverse reactions derived from previous therapies (excluding hair loss), which is over level 1 in CTC AE (5.0) abnormal blood coagulation (INR>1.5 or PT > ULN + 4s or APTT > 1.5 ULN), with bleeding tendency or receiving thrombolytic or anticoagulant therapy renal insufficiency: urinary protein ≥ ++, or 24-hour urine protein ≥ 1.0g; The effect of surgery or trauma has been eliminated for less than 14 days before enrollment Severe acute or chronic infections requiring systemic treatment Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias Patients with peripheral neuropathy which is over level 2 in CTC AE (5.0), except for trauma respiratory syndrome (dyspnea≥CTC AE 2), severe pleural effusion, ascites, pericardial effusion Long-term unhealed wounds or fractures Decompensated diabetes or other ailments treated with high doses of glucocorticoids with kinds of factors which affect oral medicine (e.g. failing to swallow, gastrointestinal tract getting resected, chronic diarrhea and ileus) hemoptysis (daily hemoptysis>50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency Thrombosis events occurring within 12 months prior to enrollment Planned to get systemic anti-tumor therapy during this study；EF-RT was performed within 4 weeks before enrollment or limited field radiotherapy within 2 weeks before grouping Hypertension (systolic blood pressure≥140 mmHg or diastolic blood pressure≥90 mmHg) that is still uncontrollable using two or more combination therapies History of psychotropic substance abuse and inability to quit or have mental disorders HIV test positive history or AIDS; untreated active hepatitis; combined with hepatitis B and hepatitis C co-infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-03-12 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
PFS（Progress free survival） | each 42 days up to PD or death (up to 24 months)
  The PFS time is defined as time from enrollment to locoregional or systemic recurrence, second malignancy or death due to any cause; censored observations will be the last date of : "death", "last tumor assessment", "last follow up date" or "last date in drug log"

SECONDARY OUTCOMES:
OS（Overall Survival） | From enrollment until death (up to 24 months)]
  OS was defined as time from date of enrollment to date of death due to any cause. For participants still alive at the time of analysis, OS time was censored on last date that participants were known to be alive.
ORR（Objective Response Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)]
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Objective Response Rate (ORR) is defined as participants who had complete response (CR) or partial response(PR) divided by the total number of patients.
DCR（Disease Control Rate） | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  To evaluate the effectiveness of Anlotinib Hydrochloric Capsule Plus Icotinib Hydrochloric Tablet by enhanced CT/MRI scan every two cycles. Disease Control Rate (DCR) defined as the percentage of participants with Disease Control best overall response (complete response, partial response or stable disease).
Adverse Events | Until 30 day safety follow-up visit
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China